CLINICAL TRIAL: NCT03485443
Title: Effects of Intraoperative Fluid Infusion on Postoperative Vomiting in Pediatric Patients Undergoing Otorhinolaryngological Surgery
Brief Title: Effects of Fluid Infusion on Postoperative Vomiting in Pediatric Patients Undergoing Otorhinolaryngological Surgery
Acronym: FLUIDVOMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Adnan Menderes University, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FLUID-VOMITING
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: fluid infusion; vomiting; otorhinolaringology
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The postoperative assessment following the anesthesiologist, nurse and parents were blind during the entire study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (%0.9 NaCl 10ml/kg) (Active Comparator): The group (Group 1) received 10 ml kg-1 throughout the entire surgical procedure.
  Four point scale using scored vomiting. m CHEOPS Scale using scored between 0-10.
  Interventions: Drug: %0.9 NaCl 10ml/kg
- Group II (%0.9 NaCl 20ml/kg) (Active Comparator): The group (Group 2) received 30 ml kg-1 throughout the entire surgical procedure.
  Four point scale using scored vomiting. m CHEOPS Scale using scored between 0-10.
  Interventions: Drug: %0.9 NaCl 20ml/kg

INTERVENTIONS:
Drug: %0.9 NaCl 10ml/kg — Fluid administration
  Arms: Group I (%0.9 NaCl 10ml/kg)
Drug: %0.9 NaCl 20ml/kg — Fluid administration
  Arms: Group II (%0.9 NaCl 20ml/kg)

SUMMARY:
Otorhinolaryngological surgery is one of the commonly applied procedures surgical treatments of children in the world. Postoperative vomiting (POV) is an important part of the management of pediatric anesthesia in this surgery that is also related with these surgical procedures. Postoperative vomiting is one of the most common complication of this surgery and may cause patients to receiving anesthesia again and stay longer in the hospital.The use of effective fluid therapy might be a safe way to reduce POV. There are many studies of fluid therapy adult patients on the other hands the number of children studies are limited.

The aim of this study was to evaluate the POV effect of intraoperative hydration with 0.9 NaCl solution in children undergoing otorhinolaryngological surgery.

DETAILED DESCRIPTION:
After institutional ethics committee approval and written informed parental consent, ASA physical status I or II, aged 2-14 year, who were undergoing elective day case otorhinolaryngological surgery under general anaesthesia, were screened for eligibility for enrollment in this prospective, randomized, double blind, placebo controlled study.

In the operating room, after routine monitoring, general anaesthesia was induced with %8 sevoflurane in 100% oxygen by a face mask with spontaneous ventilation.

Patients were randomly assigned to one of the two groups. Randomization was carried out using a computer-generated random numbers.

The control group (Group I) received ≤10 ml kg-1 h-1 and the high volüme group ( Group II) received >30 ml kg-1h-1 of intravenous %0.9 NaCl solution.Before tracheal intubation, all subjects received propofol 2:5mg kg-1, fentanyl 1µg kg-1 and rocuronium 0.6 mg kg-1.

After tracheal intubation, anaesthesia was maintained with 40% mixture of oxygen/nitrous oxide and 2% sevoflurane. The solution appears to be covered via an infusion pump was used. During anaesthesia, all patients received intravenous paracetamol 10 mg kg-1 for postoperative pain .

Following extubation, until the transfer of the patient from the time of the PACU nausea, vomiting or both were recorded..

Retching efforts in the PACU were recorded as nausea evaluated. Both nausea and vomiting were assessed on a four point scale: 0=no nausea/vomit, 1=mild nausea/vomit, patient not requesting metoclopramide, 2=nausea/vomit, patient requesting metoclopramide and 3=nausea/vomit resistant to treatment At the first episode of severely nause and vomiting, or both, a rescue antiemetic consisting of intravenous ondansetron was administered.

Intensity of pain was evaluated using Children's Hospital East Ontario Pain Scale (CHEOPS).

Knowledge collection for posoperative pain to PACU arrival and departure was performed by a postanesthesia care unit (PACU) nurses who blinded to the procedure the amount of fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* 2-14 years
* ASA I-II

Exclusion Criteria:

* Gastroesafageal reflu
* Premedication antiemetic

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
vomiting | postoperative first 30 min
  Both nausea and vomiting were assessed on a four point scale: 0=no nausea/vomit, 1=mild nausea/vomit, patient not requesting metoclopramide, 2=nausea/vomit, patient requesting metoclopramide and 3=nausea/vomit resistant to treatment

SECONDARY OUTCOMES:
Pain | postoperative first 30 min
  Intensity of pain was evaluated using Children's Hospital East Ontario Pain Scale (CHEOPS).

CONTACTS AND LOCATIONS:
Overall Officials: sinan yılmaz, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University Training and Research Hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided